CLINICAL TRIAL: NCT00434616
Title: Security and Effectiveness of Autologous Bone Marrow Stem Cell Transplantation to Avoid Amputations in Patients With Limb-threatening Ischemia: A Multicentric Randomized Placebo-controlled Double-blind Study
Brief Title: Autologous Bone Marrow Stem Cell Transplantation for Critical, Limb-threatening Ischemia
Acronym: BONMOT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Franziskus-Krankenhaus (Other)
Collaborators: Klinikum Karlsbad-Langensteinbach (Other); Stiftungsklinikum Boppard (Unknown); Krankenhaus der Barmherzigen Brüder Trier (Other)
Responsible Party: Berthold Amann, Franziskus-Krankenhaus berlin, germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-001825-24; FKH 200
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-04

CONDITIONS: Peripheral Vascular Disease; Diabetic Foot; Peripheral Arterial Occlusive Disease; Leg Ulcer; Gangrene; Ischemia
Keywords: angiogenesis; Arterial Occlusive Diseases; Leg Ulcer; Gangrene; Ischemia; PAOD; Amputation; bone marrow
MeSH Terms: conditions — Peripheral Vascular Diseases; Diabetic Foot; Peripheral Arterial Occlusive Disease 1; Leg Ulcer; Gangrene; Ischemia; Arterial Occlusive Diseases | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): saline injections
  Interventions: Biological: saline injection
- 2 (Active Comparator): autologous bone marrow transplantation into the ischemic leg
  Interventions: Procedure: Autologous bone marrow cell concentrate transplantation

INTERVENTIONS:
Procedure: Autologous bone marrow cell concentrate transplantation — bone marrow aspiration (240 ml), processing and reinjection
  Arms: 2
Biological: saline injection — saline injections
  Arms: 1

SUMMARY:
Critical limb ischemia is a condition where the blood circulation in the limbs, in most cases the legs, is decreased so that pain and non healing wounds ensue. Mostly, this is a sequel of arteriosclerosis and/or diabetes. If surgical and other methods for the improvement of blood supply for the leg have failed or are not possible, most of these patients will proceed to amputation of the leg.

Bone marrow contains cells which can induce and augment the growth of new, small arteries called collateral arteries. It has been shown in animals and in some case series that the transplantation of a concentrate of the patient's own bone marrow with stem cells into the ischemic limb can improve the blood circulation via the induction of collateral growth. However, it is not known if this bone-marrow stem cell induced collateral growth is sufficient to avoid otherwise necessary amputations.

Therefore, we conduct a study to compare the efficiency of concentrated bone marrow cells injected into the critically ischemic limb compared to a placebo procedure where only saline is injected. We think that the transplantation of autologous bone marrow will reduce the number of necessary leg amputations, reduce pain and induce wound healing. In this investigation, patients with limb threatening ischemia are randomly allocated either to the bone marrow group or to the placebo group. Patients in the bone marrow group will have their bone marrow harvested under sedation, and the bone marrow cells are concentrated. The cell concentrate will then be injected directly into the muscle of the diseased leg. Patients in the placebo group will undergo sedation as well but no bone marrow harvest is done, and saline is injected into the ischemic leg. The procedure will require about 1.5-2 hours, and the subjects will be admitted to a participating vascular Centre. Monthly examinations up to three months after the bone-marrow or placebo procedure are done. After the follow-up of three months, the rate of death and amputations and the wound healing process are compared between groups. Adverse and serious adverse events will be recorded during this time period. Diagnostic studies will be obtained to measure blood flow in the treated leg during the follow up period and include skin oxygen measurements, pressure recordings in the leg and arteriography. Also, quality of life, pain and wound healing will be assessed.

After completion of the three months study participation, subjects who have been treated with placebo will be able to receive open-label bone marrow transplantation therapy.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) represents very advanced arteriosclerosis. It is not unusual for this condition to result in limb-threatening ischemia that usually results in amputation of the limb. About 150.000 thigh or calf amputations due to PAD are done annually in the United states.

Treatment of critical limb threatening ischemia (corresponding to Rutherford grade II or III) consists of revascularization of the leg with critically reduced blood supply. Depending on the localization and morphology of the occlusion, surgical revascularization by means of bypass surgery or catheter-based percutaneous transluminal angioplasty (PTA) may be used (even as a complementary procedure). However, successful revascularization is possible in only max. 60% to 70% of the patients affected. Patients with limb threatening ischemia which cannot be revascularized have a one-year amputation rate exceeding 80% and a 20-30% mortality.

Several studies have shown that in less advanced PAD the implantation of a concentration of mononuclear cells harvested from the patient's own bone marrow has been effective in developing collateral vessel formation translating into an improvement in PAD symptoms. Additional clinical evidence that this simple, safe and inexpensive therapy can induce therapeutic angiogenesis in the ischemic limb sufficient to prevent amputation would be valuable to both patients and clinicians.

This study will evaluate the clinical potential for the implantation of a concentration of bone marrow mononuclear cells which contain stem cells for therapeutic angiogenesis through the augmented formation of collateral vessels in the ischemic limb. It is a placebo-controlled, 1:1 randomized study with a total of 90 patients included. The placebo procedure consists of a sham bone marrow puncture where no bone marrow aspiration is done; instead, only a stab puncture of the skin is made.

The bone marrow cell concentrate will be prepared "point of care", patient-side from an aspirate of 240 mL of bone marrow. A concentrate volume of 40-50 mL will be injected into 40-50 sites in the muscles of the ischemic limb. A blinded physician injects either the bone marrow cell concentrate or the visually identical placebo solution into the ischemic leg.

Improvement in perfusion of the limb will be measured using clinical assessment and ankle-brachial-index (ABI), transcutaneous oxygen (TcPO2) and contrast angiography. Quality of life and pain will be assessed.

Study participation ends for the subjects after a follow-up of three months with monthly visits. After this, clinical and perfusion status are recorded at least three-monthly up to two years after study inclusion.

HYPOTHESIS:

Implantation of Bone Marrow stem cell Aspirate Concentrate (BMAC) can be clinically effective in treating critical limb threatening ischemia so that the number of amputations can be reduced.

Inclusion criteria:

* Presence of Critical Limb ischemia according to the guidelines of the Transatlantic Consensus Group (TASC) Rutherford grade II or III. Perfusion is measured with absolute perfusion pressure and ankle-brachial index (ABI) and transcutaneous oxygen tension (TcpO2); for inclusion, ABI has to be less than or equal to 0.6 or absolute ankle pressure must be less than 60 mmHg. If ABI is technically not feasible, e.g. in patients with media calcification, inclusion criteria are a tcpO2 value (supine, forefoot, 44°C) of less than 20 mmHg if there is no tissue loss, or a tcpO2 of less than 40 mmHg if there is tissue loss.
* No sufficient response to best standard care delivered for six weeks.
* No surgical or radiological interventional option for revascularisation as confirmed by a vascular surgeon and an interventional radiologist
* Age older than 18 years
* Signed informed consent
* Absence of life-threatening complications from the ischemic limb

Exclusion criteria:

* Expected life span less than six months
* Bone marrow diseases which preclude transplantation (eg lymphoma, leukemia, myelodysplastic syndrome and others)
* Renal failure on hemodialysis
* Life threatening complications of limb ischemia with the need for immediate limb amputation to avoid death or clinical deterioration

End points:

* Primary end point: Major amputation (above the ankle) of the index limb after 3 months or persisting critical limb ischemia of the index limb after three months
* Secondary end points:

  * Wound healing (wound size, wound stage)
  * Pain and analgesics use
  * Rutherford grade and stage
  * Walking distance (treadmill) if possible
  * Quality of life (EQ-5D Questionnaire)
  * Transcutaneous oxygen pressure (TcpO2), ABI, absolute ankle perfusion pressure
  * Collateral artery number as judged by contrast angiography after 3 months
  * Rate and extent of minor (below the ankle) amputations in the index limb

ELIGIBILITY:
Inclusion Criteria:

* Presence of Critical Limb ischemia according to the guidelines of the Transatlantic Consensus Group (TASC) Rutherford grade II or III. Perfusion is measured with absolute perfusion pressure and ankle-brachial index (ABI) and transcutaneous oxygen tension (TcpO2); for inclusion, ABI has to be less than or equal to 0.6 or absolute ankle pressure must be less than 60 mmHg. If ABI is technically not feasible, e.g. in patients with media calcification, inclusion criteria are a tcpO2 value (supine, forefoot, 44°C) of less than 20 mmHg if there is no tissue loss, or a tcpO2 of less than 40 mmHg if there is tissue loss.
* No sufficient response to best standard care delivered for six weeks.
* No surgical or radiological interventional option for revascularisation as confirmed by a vascular surgeon and an interventional radiologist
* Age older than 18 years
* Signed informed consent
* Absence of life-threatening complications from the ischemic limb

Exclusion Criteria:

* Expected life span less than six months
* Bone marrow diseases which preclude transplantation (eg lymphoma, leukaemia, myelodysplastic syndrome and others)
* Renal failure on hemodialysis
* Life threatening complications of limb ischemia with the need for immediate limb amputation to avoid death or clinical deterioration

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2007-04; Primary Completion 2011-04 (Actual); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Major amputation of the index limb or persisting, unchanged critical limb ischemia | 3 months

SECONDARY OUTCOMES:
Wound healing (wound size, wound stage) | 3 months
Pain and analgesics use | 3 months
Rutherford grade and stage | 3 months
Walking distance (treadmill) if possible | 3 months
Quality of life (EQ-5D Questionnaire) | 3 months
Transcutaneous oxygen pressure (TcpO2), ABI, absolute ankle perfusion pressure | 3 months
Collateral artery number as judged by contrast angiography after 3 months | 3 months
Rate and extent of minor (below the ankle) amputations | 3 months
survival without amputation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Amann, MD, Principal Investigator — Franziskus Hospital, Berlin Vascular Center
Locations (1):
- Franziskus Hospital Berlin Vascular Center, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Tateishi-Yuyama E, Matsubara H, Murohara T, Ikeda U, Shintani S, Masaki H, Amano K, Kishimoto Y, Yoshimoto K, Akashi H, Shimada K, Iwasaka T, Imaizumi T; Therapeutic Angiogenesis using Cell Transplantation (TACT) Study Investigators. Therapeutic angiogenesis for patients with limb ischaemia by autologous transplantation of bone-marrow cells: a pilot study and a randomised controlled trial. Lancet. 2002 Aug 10;360(9331):427-35. doi: 10.1016/S0140-6736(02)09670-8. PMID 12241713
- [Background] Durdu S, Akar AR, Arat M, Sancak T, Eren NT, Ozyurda U. Autologous bone-marrow mononuclear cell implantation for patients with Rutherford grade II-III thromboangiitis obliterans. J Vasc Surg. 2006 Oct;44(4):732-9. doi: 10.1016/j.jvs.2006.06.023. Epub 2006 Aug 22. PMID 16926085
- [Background] Iba O, Matsubara H, Nozawa Y, Fujiyama S, Amano K, Mori Y, Kojima H, Iwasaka T. Angiogenesis by implantation of peripheral blood mononuclear cells and platelets into ischemic limbs. Circulation. 2002 Oct 8;106(15):2019-25. doi: 10.1161/01.cir.0000031332.45480.79. PMID 12370229 (Retraction: PMID 23704253 Circulation. 2013 Jun 11;127(23):e842)
- [Background] Nizankowski R, Petriczek T, Skotnicki A, Szczeklik A. The treatment of advanced chronic lower limb ischaemia with marrow stem cell autotransplantation. Kardiol Pol. 2005 Oct;63(4):351-60; discussion 361. English, Polish. PMID 16273471
- [Background] Hernandez P, Cortina L, Artaza H, Pol N, Lam RM, Dorticos E, Macias C, Hernandez C, del Valle L, Blanco A, Martinez A, Diaz F. Autologous bone-marrow mononuclear cell implantation in patients with severe lower limb ischaemia: a comparison of using blood cell separator and Ficoll density gradient centrifugation. Atherosclerosis. 2007 Oct;194(2):e52-6. doi: 10.1016/j.atherosclerosis.2006.08.025. Epub 2006 Sep 18. PMID 16982058
- [Background] Lawall H, Bramlage P, Amann B. Stem cell and progenitor cell therapy in peripheral artery disease. A critical appraisal. Thromb Haemost. 2010 Apr;103(4):696-709. doi: 10.1160/TH09-10-0688. Epub 2010 Feb 19. PMID 20174766
- [Background] Amann B, Luedemann C, Ratei R, Schmidt-Lucke JA. Autologous bone marrow cell transplantation increases leg perfusion and reduces amputations in patients with advanced critical limb ischemia due to peripheral artery disease. Cell Transplant. 2009;18(3):371-80. doi: 10.3727/096368909788534942. Epub 2009 Apr 2. PMID 19500466
- See also: Home page of Berlin Vascular Center — http://www.franziskus-berlin.de/